CLINICAL TRIAL: NCT00186953
Title: Determination of Optimal Dose and Safety Profile of Optison Ultrasound Contrast Agent in Pediatric Solid Tumor Patients
Brief Title: Determination of a Safe Dose of Optison in Pediatric Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPTUS
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Abdominal Neoplasms; Pelvic Neoplasms
Keywords: Ultrasound; Abdominal tumors; Pelvic tumors
MeSH Terms: conditions — Abdominal Neoplasms; Pelvic Neoplasms | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Optison

INTERVENTIONS:
Drug: Optison — Intervention description:
  Based on recommendation by the FDA, we began with a dose of 0.125ml/m^2 and escalated at 0.15 ml/m^2 increments, to 0.275 ml/m^2 and 0.425ml/m^2 and 0.500ml/m^2. We will now continue to escalate the dose of Optison at 0.300ml/m^2 increments to a maximum single dose of 4ml or a total cumulative dose of 8.7 ml as recommended by the manufacturer.

SUMMARY:
St. Jude Children's Research Hospital is studying ways to make ultrasound images clearer - to be able to see blood vessels, body structures, and tumors better. Ultrasound uses sound waves to create pictures, allowing doctors and other medical professionals to "see" inside the body.

Researchers are studying a contrast agent (like a dye) called Optison™. St. Jude Children's Research Hospital researchers want to learn the best and safest dose of this ultrasound "dye."

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-20 years old
* Subject has a known or suspected solid soft tissue tumor in the abdomen or pelvis.
* Subject is scheduled for other imaging or is already scheduled for an ultrasound or has already had adequate imaging performed at an outside institution.
* Subject is able to lie still for the exam without sedation.

Exclusion Criteria:

* Known or suspected hypersensitivity to albumin, blood or blood products.
* History of open heart surgery, cyanotic congenital heart disease or an axygen saturation of less than 96% as determined by pulse oximetry.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2002-06; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To learn the best dose of Optison™ ultrasound contrast agent that can be safely given to children with abdominal or pelvic tumors. | Unknown-study temporarily closed.
To learn the effects (good and bad) of using Optison during ultrasound. | Unknown-study temporarily closed.
To learn if using Optison™ during ultrasound can show the size and location of a tumor, how the tumor is responding to chemotherapy, and whether it has moved into surrounding tissue. | Unknown-study temporarily closed.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. McCarville, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Anderson LN, Maguire JL, Lebovic G, Hanley AJ, Hamilton J, Adeli K, McCrindle BW, Borkhoff CM, Parkin PC, Birken CS; Applied Research Group for Kids! (TARGet Kids!) Collaboration. Duration of Fasting, Serum Lipids, and Metabolic Profile in Early Childhood. J Pediatr. 2017 Jan;180:47-52.e1. doi: 10.1016/j.jpeds.2016.09.005. Epub 2016 Oct 11. PMID 27742126
- See also: St. Jude Children's Research Hospital — http://www.stjude.org